CLINICAL TRIAL: NCT03273686
Title: Efficacy of Nasogastric Tube Application in Postoperative Care of Esophagectomy: a Randomized Clinical Trial
Brief Title: Efficacy of Nasogastric Tube Application in Postoperative Care of Esophagectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiaqing Xiang, Professor of Department of Thoracic Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-NGT
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Nasogastric Tube
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group without NG tube after surgery (Experimental): In this goup, patients will undergo preoperative gastrointestinal decompression and investigators will discharge the NG tube during the surgery.
  Interventions: Procedure: Discharge the NG tube during the surgery
- group with NG tube after surgery (No Intervention): In this goup, patients will undergo preoperative gastrointestinal decompression and investigators will discharge the NG tube 6-7 days after the surgery.

INTERVENTIONS:
Procedure: Discharge the NG tube during the surgery — Discharge the NG tube during the surgery.
  Arms: group without NG tube after surgery

SUMMARY:
Nasogastric decompression is standard practice after esophageal resection in most centers because it is expected to reduce the incidence of esophagogastric anastomotic leakage by preventing overdistension of the gastric conduit. Most esophageal surgeons have been reluctant to move away from this tradition because of the considerable morbidity of anastomotic leaks after esophagectomy. However, a contrarian view is that the use of prolonged NGD may increase the incidence of postoperative pulmonary complications by promoting aspiration. Considering the numerous complications caused by using the tube and the uncertainty about its usefulness and the scarcity of studies conducted on the subject, particularly in patients with esophageal cancer, the necessity of using the tube in these types of cases is investigated in the present study.

DETAILED DESCRIPTION:
Methods In this clinical trial, patients with esophageal cancer were randomized into groups with NG tube and without NG tube after surgery. Sequence generation was performed using a computer-generated sequence of random numbers with permuted blocks. Standard postoperative management protocols were followed in both groups to avoid potential bias, which including preoperation nasogastric decompression. Thoracic esophageal mobilization and mediastinal lymphadenectomy were performed by open thoracotomy surgery. The abdominal part of the surgery was performed by laparotomy, gastric tube reconstruction was performed using linear staplers, and the conduit was brought up to the neck through the posterior mediastinal route. A cervical esophagogastric anastomosis was performed by stapled (linear) techniques. All patients were mobilized early, began early enteral feeding through jejunostomy tubes. Randomization was performed during the surgery. The group without NG tube after surgery will discharge the NG tube during the surgery. While the control group(group with NG tube after surgery) will discharge the NG tube 6-7days after surgery. The variables recorded for each patient included pulmonary complications, wound complications, anastomosis leak as well as the duration of postoperative hospitalization and the need for placing replacing the NG tube.

ELIGIBILITY:
Inclusion Criteria:

Patients who were fit for esophageal resection and underwent transthoracic or transhiatal esophagectomy with gastric tube reconstruction.

-

Exclusion Criteria:

1. Stage investigations indicating unresectable advanced disease(T4 or M1a,M1b).
2. Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment.
3. Patients with unstable situation after surgery (eg, need ventilation and ICU treatment)
4. Patients medically unfit for surgical resection.
5. Patients with pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal lymphadenectomy.
6. Mentally disabled.
7. Expected life duration of less than 3 months.
8. Patients undergoing colonic reconstruction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
postoperative complication | an expected average of 4 weeks
  the occurrence of major pulmonary complications and anastomotic leaks.

SECONDARY OUTCOMES:
the need for placing/ replacing the NG tube | an expected average of 2 weeks
  the need for placing/ replacing the NG tube
Length of postoperative stay | an expected average of 2 weeks
  Length of postoperative stay

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqing Xiang, MD, Principal Investigator — Professor of Department of Thoracic Surgery, Fudan University Shanghai Cancer Center

IPD SHARING:
Plan to Share IPD: No